CLINICAL TRIAL: NCT05255289
Title: Evaluation of Efficacy and Safety of Midurethral Slings in Women With Stress Incontinence
Brief Title: Efficacy/Safety of Midurethral Sling
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Medical College (Other)
Responsible Party: Principal Investigator, Chin-Tsung Shen, Head of administration, Mackay Medical College
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20MMHIS410e
Record Dates: First submitted 2022-02-12; First posted 2022-02-24 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (34):
- Before TOT (Experimental): Data obtained before the operation
  Interventions: Procedure: Urodynamic investigations before and after a trans-obturator tape protocol.
- After TOT (Experimental): Data obtained after the operation
  Interventions: Procedure: Urodynamic investigations before and after a trans-obturator tape protocol.
- Before TVT-O (Experimental): Data obtained before the operation.
  Interventions: Procedure: Urodynamic investigations before and after a tension-free vaginal tape-obturator (TVT-O)
- After TVT-O (Experimental): Data obtained after the operation.
  Interventions: Procedure: Urodynamic investigations before and after a tension-free vaginal tape-obturator (TVT-O)
- Aged patient (>50 y/o) before TVT-O (Experimental): Data obtained before the operation.
  Interventions: Procedure: Urodynamic investigations before and after a tension-free vaginal tape-obturator (TVT-O)
- Aged patient (>50 y/o) after TVT-O (Experimental): Data obtained after the operation.
  Interventions: Procedure: Urodynamic investigations before and after a tension-free vaginal tape-obturator (TVT-O)
- Young patients (<50 y/o) before TVT-O (Experimental): Data obtained before the operation.
  Interventions: Procedure: Urodynamic investigations before and after a tension-free vaginal tape-obturator (TVT-O)
- Young patients (<50 y/o) after TVT-O (Experimental): Data obtained after the operation.
  Interventions: Procedure: Urodynamic investigations before and after a tension-free vaginal tape-obturator (TVT-O)
- Menopausal patient before TVT-O (Experimental): Data obtained before the operation.
  Interventions: Procedure: Urodynamic investigations before and after a tension-free vaginal tape-obturator (TVT-O)
- Menopausal patient after TVT-O (Experimental): Data obtained after the operation.
  Interventions: Procedure: Urodynamic investigations before and after a tension-free vaginal tape-obturator (TVT-O)
- Pre-menopausal patient before TVT-O (Experimental): Data obtained before the operation.
  Interventions: Procedure: Urodynamic investigations before and after a tension-free vaginal tape-obturator (TVT-O)
- Pre-menopausal patients after TVT-O (Experimental): Data obtained after the operation.
  Interventions: Procedure: Urodynamic investigations before and after a tension-free vaginal tape-obturator (TVT-O)
- Before i-STOP (Experimental): Data obtained before the operation.
  Interventions: Procedure: Urodynamic investigations before and after an i-STOP mini adjustable sling protocol.
- After i-STOP (Experimental): Data obtained after the operation.
  Interventions: Procedure: Urodynamic investigations before and after an i-STOP mini adjustable sling protocol.
- Aged patient before i-STOP (Experimental): Data obtained before the operation.
  Interventions: Procedure: Urodynamic investigations before and after an i-STOP mini adjustable sling protocol.
- Aged patient after i-STOP (Experimental): Data obtained after the operation.
  Interventions: Procedure: Urodynamic investigations before and after an i-STOP mini adjustable sling protocol.
- Young patient before i-STOP (Experimental): Data obtained before the operation.
  Interventions: Procedure: Urodynamic investigations before and after an i-STOP mini adjustable sling protocol.
- Young patient after i-STOP (Experimental): Data obtained after the operation.
  Interventions: Procedure: Urodynamic investigations before and after an i-STOP mini adjustable sling protocol.
- Menopausal patient before i-STOP (Experimental): Data obtained before the operation.
  Interventions: Procedure: Urodynamic investigations before and after an i-STOP mini adjustable sling protocol.
- Menopausal patient after i-STOP (Experimental): Data obtained after the operation.
  Interventions: Procedure: Urodynamic investigations before and after an i-STOP mini adjustable sling protocol.
- Pre-menopausal patient before i-STOP (Experimental): Data obtained before the operation.
  Interventions: Procedure: Urodynamic investigations before and after an i-STOP mini adjustable sling protocol.
- Pre-menopausal patient after i-STOP (Experimental): Data obtained after the operation.
  Interventions: Procedure: Urodynamic investigations before and after an i-STOP mini adjustable sling protocol.
- Before mini Arc (Experimental): Data obtained before the operation.
  Interventions: Procedure: Urodynamic investigations before and after a mini Arc protocol.
- After mini Arc (Experimental): Data obtained after the operation.
  Interventions: Procedure: Urodynamic investigations before and after a mini Arc protocol.
- Age patient before mini Arc (Experimental): Data obtained before the operation.
  Interventions: Procedure: Urodynamic investigations before and after a mini Arc protocol.
- Age patient after mini Arc (Experimental): Data obtained after the operation.
  Interventions: Procedure: Urodynamic investigations before and after a mini Arc protocol.
- Young before mini Arc (Experimental): Data obtained before the operation.
  Interventions: Procedure: Urodynamic investigations before and after a mini Arc protocol.
- Young patient after mini Arc (Experimental): Data obtained after the operation.
  Interventions: Procedure: Urodynamic investigations before and after a mini Arc protocol.
- Menopausal patient before mini Arc (Experimental): Data obtained before the operation.
  Interventions: Procedure: Urodynamic investigations before and after a mini Arc protocol.
- Menopausal patient after mini Arc (Experimental): Data obtained after the operation.
  Interventions: Procedure: Urodynamic investigations before and after a mini Arc protocol.
- Pre-menopausal before mini Arc (Experimental): Data obtained before the operation.
  Interventions: Procedure: Urodynamic investigations before and after a mini Arc protocol.
- Pre-menopausal patient after mini Arc (Experimental): Data obtained after the operation.
  Interventions: Procedure: Urodynamic investigations before and after a mini Arc protocol.
- Before Solyx sling (Experimental): Data obtained before the operation
  Interventions: Procedure: Urodynamic investigations before and after an Solyx sling protocol.
- After Solyx sling (Experimental): Data obtained before the operation
  Interventions: Procedure: Urodynamic investigations before and after an Solyx sling protocol.

INTERVENTIONS:
Procedure: Urodynamic investigations before and after a trans-obturator tape protocol. — Urodynamic investigations (The urodynamic study included free uroflowmetry, postvoid residual, filling and voiding cystometry, and a urethral pressure profile. The filling cystometry and urethral pressure profile were performed with 37 degrees C normal saline similar to body temperature at an infusion rate of 80 ml/min.)
  Arms: After TOT; Before TOT
Procedure: Urodynamic investigations before and after a tension-free vaginal tape-obturator (TVT-O) — Urodynamic investigations (stated above.)
  Arms: After TVT-O; Aged patient (>50 y/o) after TVT-O; Aged patient (>50 y/o) before TVT-O; Before TVT-O; Menopausal patient after TVT-O; Menopausal patient before TVT-O; Pre-menopausal patient before TVT-O; Pre-menopausal patients after TVT-O; Young patients (<50 y/o) after TVT-O; Young patients (<50 y/o) before TVT-O
Procedure: Urodynamic investigations before and after a mini Arc protocol. — Urodynamic investigations (stated above)
  Arms: After mini Arc; Age patient after mini Arc; Age patient before mini Arc; Before mini Arc; Menopausal patient after mini Arc; Menopausal patient before mini Arc; Pre-menopausal before mini Arc; Pre-menopausal patient after mini Arc; Young before mini Arc; Young patient after mini Arc
Procedure: Urodynamic investigations before and after an i-STOP mini adjustable sling protocol. — Urodynamic investigations (stated above)
  Arms: After i-STOP; Aged patient after i-STOP; Aged patient before i-STOP; Before i-STOP; Menopausal patient after i-STOP; Menopausal patient before i-STOP; Pre-menopausal patient after i-STOP; Pre-menopausal patient before i-STOP; Young patient after i-STOP; Young patient before i-STOP
Procedure: Urodynamic investigations before and after an Solyx sling protocol. — Urodynamic investigations (stated above.)
  Arms: After Solyx sling; Before Solyx sling

SUMMARY:
The trans-obturator tape (TOT), which exhibits a satisfactory cure rate and a relatively diminished invasiveness, has been increasingly accepted as a surgical treatment of stress urinary incontinence (SUI) patients. Nevertheless, in contrast to the well-recognized therapeutic benefit of the enhanced resistance to the bladder continence during urine storage, if the voiding function of the bladder adapts to the TOT-enhanced outlet resistance has not been adequately investigated. This study retrospectively assayed the voiding efficacy of each voiding cycle, to clarify if the thermodynamic efficacy of the bladder was modified in response to the TOT surgery.

DETAILED DESCRIPTION:
The urodynamic study included free uroflowmetry, postvoid residual, filling and voiding cystometry, and a urethral pressure profile. The filling cystometry and urethral pressure profile were performed with 37 degrees C normal saline similar to body temperature at an infusion rate of 80 ml/min. All patients received a pre- and a post-operative urodynamic evaluation, in which pre-operative evaluation was conducted 1-4 weeks before TOT procedure, and post-operative evaluation was done at 4-6 weeks follow-up.

Complete multichannel urodynamic studies including free uroflowmetry, filling and voiding cystometry, and urethral pressure profile was performed in each patient. The urodynamic parameters measured were the maximum flow rate (Qmax), voided volume, post-void residual volume (PVR), and detrusor pressure at Qmax (Pdet. Qmax). The filling cystometry and urethral pressure profile were performed with 37 degrees C normal saline at an infusion rate of 80 ml/min. All data were recorded and analyzed using a Medical Measurement Systems (MMS UD-200, Enschede, The Netherlands). All data in this study will be expressed as mean ± SEM. After checking the normality and variance of data, two-way ANOVAs were used to assess the difference in values among testing groups and time points; and post hoc Student-Newman-Keuls tests were used to compare the means of groups when there was a significant difference between groups. Significance was set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stress urinary incontience
* Have urodynamic investigations before and after operation.

Exclusion Criteria:

* Exclusion criteria will be a history of (1) cardiovascular, (2) neurological, or (3) other medical (such as diabetes or inflammation) problems as well as (4) patients who received a concomitant surgical procedure.

Ages: 30 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Pressure-volume study | within a voiding cycle (a cycle is about 30 to 60 minutes)
  urine leakage.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Shing Leu, M.D., Study Chair — Department of Ear, Nose, and Throat, MacKay Memorial Hospital, Taipei, Taiwan
Locations (1):
- Department of Obstetrics and Gynecology, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
For we uncertain if this might violate personal information laws in our country.

REFERENCES:
- [Background] Abrams P, Andersson KE, Apostolidis A, Birder L, Bliss D, Brubaker L, Cardozo L, Castro-Diaz D, O'Connell PR, Cottenden A, Cotterill N, de Ridder D, Dmochowski R, Dumoulin C, Fader M, Fry C, Goldman H, Hanno P, Homma Y, Khullar V, Maher C, Milsom I, Newman D, Nijman RJM, Rademakers K, Robinson D, Rosier P, Rovner E, Salvatore S, Takeda M, Wagg A, Wagner T, Wein A; members of the committees. 6th International Consultation on Incontinence. Recommendations of the International Scientific Committee: EVALUATION AND TREATMENT OF URINARY INCONTINENCE, PELVIC ORGAN PROLAPSE AND FAECAL INCONTINENCE. Neurourol Urodyn. 2018 Sep;37(7):2271-2272. doi: 10.1002/nau.23551. Epub 2018 Aug 14. No abstract available. PMID 30106223
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-committee of the International Continence Society. The standardisation of terminology of lower urinary tract function: report from the Standardisation Sub-committee of the International Continence Society. Neurourol Urodyn. 2002;21(2):167-78. doi: 10.1002/nau.10052. No abstract available. PMID 11857671
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, Van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-Committee of the International Continence Society. The standardisation of terminology in lower urinary tract function: report from the standardisation sub-committee of the International Continence Society. Urology. 2003 Jan;61(1):37-49. doi: 10.1016/s0090-4295(02)02243-4. No abstract available. PMID 12559262
- [Background] Atis G, Arisan S, Ozagari A, Caskurlu T, Dalkilinc A, Ergenekon E. Tissue reaction of the rat urinary bladder to synthetic mesh materials. ScientificWorldJournal. 2009 Oct 2;9:1046-51. doi: 10.1100/tsw.2009.120. PMID 19802500
- [Background] de Leval J. Novel surgical technique for the treatment of female stress urinary incontinence: transobturator vaginal tape inside-out. Eur Urol. 2003 Dec;44(6):724-30. doi: 10.1016/j.eururo.2003.09.003. PMID 14644127
- [Background] Hsiao SM, Kuo HC. Predictors of further anti-incontinence interventions or transvaginal urethrolysis after a pubovaginal sling procedure in women with and without neurologic disorders. J Formos Med Assoc. 2021 Jul;120(7):1464-1477. doi: 10.1016/j.jfma.2020.12.029. Epub 2021 Jan 16. PMID 33468403
- [Background] Huang WC, Lau HH, Su TH. Did surgical failure and complications affect incontinence-related quality of life in women after transobturator sling procedure? Taiwan J Obstet Gynecol. 2018 Apr;57(2):295-299. doi: 10.1016/j.tjog.2018.02.020. PMID 29673676
- [Background] Medina CA, Costantini E, Petri E, Mourad S, Singla A, Rodriguez-Colorado S, Ortiz OC, Doumouchtsis SK. Evaluation and surgery for stress urinary incontinence: A FIGO working group report. Neurourol Urodyn. 2017 Feb;36(2):518-528. doi: 10.1002/nau.22960. Epub 2016 Mar 7. PMID 26950893
- [Background] Schimpf MO, Rahn DD, Wheeler TL, Patel M, White AB, Orejuela FJ, El-Nashar SA, Margulies RU, Gleason JL, Aschkenazi SO, Mamik MM, Ward RM, Balk EM, Sung VW; Society of Gynecologic Surgeons Systematic Review Group. Sling surgery for stress urinary incontinence in women: a systematic review and metaanalysis. Am J Obstet Gynecol. 2014 Jul;211(1):71.e1-71.e27. doi: 10.1016/j.ajog.2014.01.030. Epub 2014 Jan 30. PMID 24487005
- [Background] Ulmsten U, Henriksson L, Johnson P, Varhos G. An ambulatory surgical procedure under local anesthesia for treatment of female urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 1996;7(2):81-5; discussion 85-6. doi: 10.1007/BF01902378. PMID 8798092
- [Background] Waltregny D, Gaspar Y, Reul O, Hamida W, Bonnet P, de Leval J. TVT-O for the treatment of female stress urinary incontinence: results of a prospective study after a 3-year minimum follow-up. Eur Urol. 2008 Feb;53(2):401-8. doi: 10.1016/j.eururo.2007.08.021. Epub 2007 Aug 21. PMID 17728052
- [Derived] Lau HH, Lai CY, Peng HY, Hsieh MC, Su TH, Lee JJ, Lin TB. Modification of bladder thermodynamics in stress urinary incontinence patients submitted to trans-obturator tape: A retrospective study based on urodynamic assessment. Front Bioeng Biotechnol. 2022 Aug 19;10:912602. doi: 10.3389/fbioe.2022.912602. eCollection 2022. PMID 36061421
- See also: Reported complications of tension-free vaginal tape procedures: A review — https://bcmj.org/sites/default/files/public/BCMJ_49_Vol9_articles_reported_complications.pdf